CLINICAL TRIAL: NCT04238403
Title: Peer Professionals to Increase Capacity to Treat ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York University (Other)
Responsible Party: Principal Investigator, Dr. Anil Chacko, Principal Investigator, New York University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FY20203646
Record Dates: First submitted 2019-12-18; First posted 2020-01-23 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Attention Deficit and Disruptive Behavior Disorders
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Parent Training (Experimental): Parent training intervention based on social learning and operant conditioning theory, generally referred to as Behavioral Parent Training.
  Interventions: Behavioral: Behavioral Parent Training (MATCH Protocol)

INTERVENTIONS:
Behavioral: Behavioral Parent Training (MATCH Protocol) — BPT. Behavioral Parent Training (BPT) is a well-established psychosocial intervention for the treatment for ADHD and related behavioral difficulties (e.g., oppositional problems). BPT is based on social learning and operant conditioning principles in which parents are instructed to utilize methods (e.g., praise, effective communication, reward systems, time-out from positive reinforcement) to facilitate positive behaviors in their child (e.g., compliance) and reduce challenging behaviors (e.g., opposition). BPT comes in several manualized, commercially available manuals. The version of BPT that we will be utilizing is from the MATCH protocol (Chorpita and Weisz, 2009), which consists of 10 components, delivered with individual families, typically over the course of 10-16 weekly individual meetings (total meetings depends upon parent availability and acquisition of BPT skills).

SUMMARY:
The goal of this 1-year project is to evaluate a service delivery model by peer support organizations to increase mental health service access and utilization for children at risk for attention-deficit/hyperactivity disorder (ADHD) from socioeconomically disadvantaged, urban communities. Behavioral parent training [BPT] currently delivered directly by Family Peer Advocates (FPAs), will be evaluated in a sample of 18 families on child outcomes.

DETAILED DESCRIPTION:
The goal of this 1-year project is to further refine and evaluate an existing and employed potentially highly sustainable and scalable service delivery model that leverages peer support organizations to increase mental health service access and utilization for children at risk for attention-deficit/hyperactivity disorder (ADHD) from socioeconomically disadvantaged, urban communities by improving the delivery of an evidence-based treatment (i.e., behavioral parent training [BPT]) currently delivered directly by Family Peer Advocates (FPAs) to parents of these children. Specifically, through an iterative, single-case cohort design, the investigators will work with FPAs to iteratively refine an existing and employed intervention model with three cohorts of parents (n= 6 families/cohort over 3 cohorts with a total sample size of 18 families). the investigators will collect information from parents before, during and after BPT to assess the impact of BPT on parents perceptions of their child's behavior and functioning, and parenting factors (e.g., parenting behavior, stress, depressive symptoms). In addition, the investigators will utilize this project to gain a better understanding of how best the position the FPA ADHD Model within the broader service delivery system through qualitative interviews with these parents to assess their experience and insights into improving the model. This research project is an effort at evaluating an existing intervention model and refining it through an iterative process.

ELIGIBILITY:
Inclusion Criteria:

* being a parent of a child who is seeking services through a participating Vibrant Emotional Health site
* being an adult over the age of 18
* having a child between the age of 5-12
* parent must speak English, Spanish, Mandarin, and/or Cantonese.

Exclusion Criteria:

• parent presenting with severe mental health illness (e.g., schizophrenia; bipolar disorder) that would warrant immediate services.

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in Impairment Rating Scale (IRS) immediately after the intervention | Assessing change from start of intervention through end of intervention at 10 weeks
  Parent report on 6 point likert scale (scores 1-6 with lower scores equating to less impairment) assessing impairment associated with children's symptoms on academic, parent, family, functioning

SECONDARY OUTCOMES:
Change in Parenting Sense of Competence Scale (PSOC) immediately after the intervention | Assessing change from start of intervention through end of intervention at 10 weeks
  The Parenting Sense of Competence Scale (PSOC) is an often used scale to assess parental competence in child-rearing. The PSOC has two factors: parenting efficacy and satisfaction and a total sum score for total parenting sense of competence. Seventeen items are rated on a 1 (strongly disagree) to 6 (strongly agree) scale. Higher scores equate to greater sense of parenting competence.
Change in Alabama Parenting Questionnaire- Short Form (APQ-SF) immediately after the intervention | Assessing change from start of intervention through end of intervention at 10 weeks
  The Alabama Parenting Questionnaire- Short Form (APQ-SF) is a well-validated 9- item measure of parenting style. Items are rated by the parent scored based on frequency of parenting behavior from Never (1), Almost Never (2), Sometimes (3), Often (4), Always (5). APQ-SF items are based around the three main structures: positive parenting, inconsistent discipline and poor supervision. Higher scores equate to better parenting skills.
Change in Beck Depression Inventory-II immediately after the intervention | Assessing change from start of intervention through end of intervention at 10 weeks
  The Beck Depression Inventory-II (BDI-II; Beck & Steer; 1987; Beck, Ward, Mendelsohn, Mock, & Erbaugh, 1961) is a 21-item self-report measure used to assess maternal depressive symptoms. Mothers were instructed to indicate which of four statements best described how they felt over the preceding two week period. The BDI is scored from one to four, with higher scores on the BDI indicating a greater degree of depression. A total score on the BDI, which is a sum of the 21-item measure, will be used in the study.
Change in Parental Stress-Short Form (PSI-SF) immediately after the intervention | Assessing change from start of intervention through end of intervention at 10 weeks
  The Parental Stress-Short Form (PSI-SF) is a 36-item self-report measure used to assess parenting stress in three domains, Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. The PSI-SF is measured along a 5-point scale with one (Strongly Disagree) to five (Strongly Agree). Higher scores indicate greater levels of parenting stress. For this study, the Total Stress score, which is the sum of the three PSI-SF domains, will be used.
Change in IOWA immediately after the intervention Connors Rating Scale (IOWA-CRS) | Assessing change from start of intervention through end of intervention at 10 weeks
  ADHD and oppositional behavior will be measured by the IOWA Connors Rating Scale (IOWA-CRS)-. The IOWA-CRS (Waschbusch & Willoughby, 2008) is a widely used brief measure of attention-deficit/hyperactivity disorder and oppositional-defiant behavior in children completed by parents. The IOWA-CRS consists of 10 items evaluated using a four-point Likert scale with the following anchors: not at all (0); just a little (1); pretty much (2); and very much (3). Higher scores equates to higher severity of behavior problems

CONTACTS AND LOCATIONS:
Overall Officials: Anil Chacko, PhD, Principal Investigator — New York University
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No